CLINICAL TRIAL: NCT04527601
Title: Extremely Premature Births During the Peak of the COVID-19 Pandemic: an International Study of the Active SafeBoosC III Departments
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Gorm Greisen, MD, professor, Rigshospitalet, Denmark
Other Study IDs: SafeBoosC COVID-19 ELGAN study
Record Dates: First submitted 2020-08-25; First posted 2020-08-26 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Extreme Prematurity; Covid19
Keywords: extreme prematurity; safeboosc; RCT; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ELGAN admissions during peak three months of COVID-19 pandemic
- ELGAN admissions in the three corresponding months of 2019

SUMMARY:
This is a retrospective, observational study based on the consortium of the SafeBoosC-III randomised clinical trial. This study will evaluate if the number of admitted extremely preterm infants has decreased in the SafeBoosC-III departments during the global lockdown, and whether there is an association between the level of lockdown restrictions and change in the number of ELGAN admissions.

DETAILED DESCRIPTION:
On the 11th of March 2020, COVID-19 was declared a pandemic by the World Health Organisation, which led to an almost worldwide lockdown (1). During the lockdown, reductions in preterm birth rates and very low birth weight infants have been reported in both Danish and Irish studies. Within the SafeBoosC-III investigator group, several neonatologists concurrently observed that the number of extremely low gestational age neonates (ELGAN) (gestational age below 28 weeks) admitted to their respective departments, had declined during the pandemic, while others observed no difference in the number of admitted ELGAN (oral communication). Furthermore, despite a 60% increase in the number of hospitals open for randomisation in the SafeBoosC-III trial from January to May, the randomisation rate has not increased as expected. Investigators are therefore curious to evaluate if the number of admitted extremely preterm infants has decreased in the SafeBoosC-III departments during the global lockdown, and whether there is an association between the level of lockdown restrictions and change in the number of ELGAN admissions. Investigators hope that this study will contribute further to the knowledge of the COVID-19 pandemics' effect on ELGAN birth as well as its effect on international randomised clinical trials.

This is a retrospective, observational study based on the consortium of the SafeBoosC-III randomised clinical trial. The SafeBoosC-III trial investigates the benefit and harms of treatment guided by cerebral near-infrared spectroscopy monitoring compared with treatment and monitoring as usual in extremely preterm infants. All 79 neonatal intensive care units (NICU) that are active in the consortium will be invited to participate in this study. Primary investigators will be contacted and asked to provide the number of extremely low gestational age neonates (ELGAN) admitted to their NICU within the most rigorous three months of the COVID-19 pandemic as well as the number of ELGAN admitted within the same period in 2019. The most rigorous three months of the COVID-19 pandemic will be a subjective definition by the local investigator, based on when the lockdown restrictions were strictest. Investigators will be asked to clarify how and where the information has been obtained from. Furthermore, investigators will be asked to classify the level of restrictions imposed upon the public, during the lockdown period, in a Likert scale format from 1-5. Additionally, investigators will be asked to categorize the impact of the COVID-19 lockdown on the everyday life of a pregnant woman.

The number of ELGAN admissions during the three peak months in total, during the same months in 2019, within each region and within each level of lockdown restriction, will be reported as numbers. The primary outcome and the secondary outcome regarding the difference in the number of ELGAN admissions between years and regions will be analysed by using Fisher's Exact test for 1x2 tables. To analyse the correlation between the level of lockdown restrictions and the change in number of ELGAN admissions, investigators will use simple linear regression. The exploratory outcome investigating if lockdown restrictions could lead to non-admittance of ELGAN will not undergo statistical analysis but will be reported and discussed. For the primary outcome, an alfa level of 5% is chosen as a threshold for significance. To correct for multiple testing in the secondary outcomes, investigators have chosen an alfa level of 1%

In a previous funding application for the SafeBoosC-III trial, investigators estimated that the 93 departments taking part in the application, had a total of 3000 ELGAN admissions per year. Therefore, investigators expect participating departments on average to have had approximately 30 admissions in 2019, i.e. approximately seven admissions in a three months period. Therefore, if half of the NICUs (i.e. 40 departments) participate, investigators would expect a total of 280 EP infant admissions within the 40 departments in 2019. Thus, a 16.5% change in the primary outcome is needed to show a statistical significance at a 5% alfa level.

ELIGIBILITY:
Inclusion Criteria:

* Extremely low gestational age neonates admitted to participating NICUs

Exclusion Criteria:

-

Ages: 22 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extremely premature infants (GA<28)
Sampling Method: Non-Probability Sample
Enrollment: 885 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
Number of ELGAN admissions during peak three months of COVID-19 compared to corresponding months in 2019 | 3 months
  The primary outcome will be the difference in the total number of ELGAN admissions in SafeBoosC-III departments during the peak three months of the COVID-19 pandemic in 2020 compared to the same three months period in 2019. The most rigorous three months of the COVID-19 pandemic will be a subjective definition by the local investigator, based on when the lockdown restrictions were strictest.

SECONDARY OUTCOMES:
Regional difference in ELGAN admissions during peak three months of COVID-19 compared to corresponding months in 2019 | 3 months
  The difference in the number of ELGAN admissions during the peak three months of the COVID-19 pandemic versus the same three months in 2019, within the following regions:
  North America: USA Northern Europe: Denmark, Norway Eastern Europe: Austria, Poland, Czech Republic, Ukraine, Turkey Western Europe: Germany, UK, Ireland, Switzerland, Belgium Southern Europe: Spain, Portugal, Italy, Greece Asia: India, China
Correlation between the level of lockdown restrictions and number of ELGAN admissions during peak three months of COVID-19 compared to corresponding months in 2019 | 3 months
  Investigators will be asked to clarify how and where the information has been obtained from. Furthermore, investigators will be asked to classify the level of restrictions imposed upon the public, during the lockdown period, in a Likert scale format from 1-5.

OTHER OUTCOMES:
Likelihood of restrictions leading to non-admittance of ELGAN | 3 months
  For the purpose of an exploratory analysis, we will ask investigators to rate the likelihood that restrictions outside or inside health institutions in their country/region, have led to non-admittance of ELGAN. Causes could be intrauterine death, or no transfer from place of birth

CONTACTS AND LOCATIONS:
Overall Officials: Gorm Greisen, MD, Prof, Study Director — Rigshospitalet, Denmark
Locations (1):
- Neonatalklinikken, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen ML, Pellicer A, Gluud C, Dempsey E, Mintzer J, Hyttel-Sorensen S, Heuchan AM, Hagmann C, Ergenekon E, Dimitriou G, Pichler G, Naulaers G, Cheng G, Guimaraes H, Tkaczyk J, Kreutzer KB, Fumagalli M, Claris O, Lemmers P, Fredly S, Szczapa T, Austin T, Jakobsen JC, Greisen G. Cerebral near-infrared spectroscopy monitoring versus treatment as usual for extremely preterm infants: a protocol for the SafeBoosC randomised clinical phase III trial. Trials. 2019 Dec 30;20(1):811. doi: 10.1186/s13063-019-3955-6. PMID 31888764
- [Derived] Rasmussen MI, Hansen ML, Pichler G, Dempsey E, Pellicer A, El-Khuffash A, A S, Piris-Borregas S, Alsina M, Cetinkaya M, Chalak L, Ozkan H, Baserga M, Sirc J, Fuchs H, Ergenekon E, Arruza L, Mathur A, Stocker M, Otero Vaccarello O, Szczapa T, Sarafidis K, Krolak-Olejnik B, Memisoglu A, Reigstad H, Rafinska-Wazny E, Hatzidaki E, Peng Z, Gkentzi D, Viellevoye R, De Buyst J, Mastretta E, Wang P, Hahn GH, Bender L, Cornette L, Tkaczyk J, Del Rio R, Fumagalli M, Papathoma E, Wilinska M, Naulaers G, Sadowska-Krawczenko I, Lecart C, Couce ML, Fredly S, Heuchan AM, Karen T, Greisen G. Extremely Preterm Infant Admissions Within the SafeBoosC-III Consortium During the COVID-19 Lockdown. Front Pediatr. 2021 Jul 12;9:647880. doi: 10.3389/fped.2021.647880. eCollection 2021. PMID 34322460
- See also: trial website — http://www.safeboosc.eu